CLINICAL TRIAL: NCT04333316
Title: Principal Investigator
Brief Title: Dual Mobility Cup: Does it Improve Patient's Satisfaction After Total Hip Arthroplastry?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, ahmed m. samy, assistant professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 42687
Record Dates: First submitted 2020-03-30; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Patient Satisfaction; Hip Osteoarthritis
Keywords: hip arthroplasty; satisfaction; dual mobility cup
MeSH Terms: conditions — Patient Satisfaction; Osteoarthritis, Hip; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This is prospective study was carried out on 180 patients with a unilateral arthritic hip between January 2011 and August 2018. Patients were divided into two groups, each group included 90 patients. Group A included patients received total hip with a large head (32-36mm.) made of cobalt-chrome. The femoral component was a cementless porous coated stem. The cup was a cementless porous coated Trilogy cup and was inserted press fit with primary additional one to three screws. Group B included those received total hip with a dual mobility cup
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- large head group (Other): study the postoperative patient's satisfaction
  Interventions: Procedure: large head; Procedure: dual mobility cup
- dual mobility group (Other): study the postoperative patient's satisfaction
  Interventions: Procedure: large head; Procedure: dual mobility cup

INTERVENTIONS:
Procedure: large head — implantation of large head total hip
Procedure: dual mobility cup — implantation of dual mobility total hip

SUMMARY:
Although the success of total hip arthroplasty, many patients were dissatisfied postoperatively. Patient's reported outcome measures become of a great importance in assessment of the results after joint replacement. The aim of this prospective study is to evaluate and compare postoperative patient's satisfaction after implantation of two commonly used different designs of total hip arthroplasty.

DETAILED DESCRIPTION:
The investigators conducted a prospective comparative study carried out on 180 patients suffering of hip arthritis between 2011 and 2018. They were randomized into two groups of homogenous demographic and clinical data. Group A was treated by cementless T.H.A. with a large head while group B received cementless T.H.A. with a dual mobility cup. Clinical evaluation and preoperative patient's expectation were assessed and compared to the postoperative satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral hip arthritis
* Age up to 65 years
* Body mass index (BMI) up to 35
* Modified Charnley comorbidity classification equal to A

Exclusion Criteria:

* Neurological deficit (e.g. Parkinsonism, stroke)
* Bone type c not fit for cementless fixation
* Poly-arthritis, active inflammatory arthritis (e.g. rheumatoid arthritis)
* Any patient with psychiatric disorders

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
patient's satisfaction | about 5 years
  measurement by patient's reported outcomes measures
clinical evaluation | about 5 years
  WOMAC score
pain assessment | about 5 years
  VAS score

IPD SHARING:
Plan to Share IPD: No
We conducted a prospective comparative study carried out on 180 patients suffering of hip arthritis between 2011 and 2018. They were randomized into two groups of homogenous demographic and clinical data. Group A was treated by cementless T.H.A. with a large head while group B received cementless T.H.A. with a dual mobility cup. Clinical evaluation and preoperative patient's expectation were assessed and compared to the postoperative satisfaction

REFERENCES:
- [Derived] Samy AM, Mahmoud AA, El-Tantawy A. Dual Mobility Cup: Does It Improve Patient's Satisfaction After Total Hip Arthroplasty? A Prospective Comparative Randomized Study. J Am Acad Orthop Surg. 2021 Nov 15;29(22):e1141-e1150. doi: 10.5435/JAAOS-D-20-00882. PMID 33252552